CLINICAL TRIAL: NCT06671574
Title: Emotional Intelligence and Relaxation Techniques in Mental Health, Sleep Disorders, and Quality of Life in Adults Over 60 Years
Brief Title: Emotional Intelligence and Relaxation Techniques for Mental Health and Sleep in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ^University of Jaén^
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Older People
MeSH Terms: interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This group will not receive intervention, but will receive information sessions on general health and well-being topics, such as sleep hygiene, healthy lifestyle habits and practical tips to improve rest, in order to control for the placebo effect. These information sessions will be held at the beginning of the study and will be supported by brochures and educational material.
- Experimental Group (Experimental): This group will participate in a structured program that combines the development of emotional intelligence with relaxation techniques. It will last 12 weeks, with sessions twice a week, each lasting approximately 60 minutes. The sessions will be led by a mental health professional. During the sessions, exercises will be worked on to recognize, understand and regulate emotions, allowing participants to develop skills to better manage stress and anxiety. In addition, relaxation techniques such as deep breathing, guided meditation and visualization will be practiced, which have been shown to be effective in reducing muscle tension, lowering cortisol levels and promoting restful sleep.
  Interventions: Other: Emotional intelligence and Relaxation techniques

INTERVENTIONS:
Other: Emotional intelligence and Relaxation techniques — In each session, participants will engage in exercises aimed at recognizing, understanding, and regulating their emotions. These interactive activities will foster personal reflection and group discussion, helping individuals identify emotions in various situations and their impact on behavior. This approach will enhance emotional awareness and equip participants with practical tools for managing stress and anxiety. Various relaxation techniques will also be introduced. Deep breathing exercises will teach participants to calm their minds and bodies, reducing tension. Guided meditation will help them focus inward, promoting mental peace and deep relaxation. Additionally, visualization exercises will encourage imagining calming scenarios, alleviating anxiety and improving overall well-being.
  Arms: Experimental Group

SUMMARY:
This topic highlights the role of emotional intelligence and relaxation techniques in enhancing mental health for adults over 60. Emotional intelligence, which involves understanding and managing one's emotions, can improve emotional well-being in older adults facing challenges like loneliness and anxiety. Sleep disorders are common in this age group and can lead to increased mental health issues such as depression. Relaxation techniques, including meditation, yoga, and deep breathing, have been shown to reduce stress and improve sleep quality. By integrating emotional intelligence and relaxation practices into daily life, older adults can enhance their overall quality of life and mental health.

ELIGIBILITY:
Inclusion Criteria:

* People aged 60 years or older.
* Older adults with mental health problems, such as anxiety, stress, or mild depressive symptoms.
* Participants who report difficulty falling or staying asleep, or who have some type of sleep disorder (such as insomnia or fragmented sleep).
* People willing to participate in emotional intelligence interventions and relaxation techniques.
* Older adults who live in a stable environment (private housing, community centers, etc.) and who have sufficient cognitive abilities to understand and follow basic instructions for relaxation techniques.

Exclusion Criteria:

* People under 60 years of age.
* Older adults with serious psychiatric disorders, such as advanced dementia, schizophrenia, or uncontrolled bipolar disorder, that could interfere with effective participation in the interventions.
* Participants with serious physical health problems, such as unstable heart disease or advanced respiratory failure, that could be worsened by relaxation techniques or limit their participation.
* People who are already receiving specific treatment for sleep disorders that includes medication or intensive psychotherapeutic interventions, since these could interfere with the results of the study.
* Older adults with severe sensory limitations (such as deafness or uncorrected blindness) that prevent them from understanding or adequately performing the proposed relaxation techniques.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
The Short Form-36 Health Survey (SF-36) | Up to twelve weeks
  Used extensively for assessing health-related quality of life. The results are values between 0 and 100. Optimal health is represented by scores of 100 and very poor health would equal 0.
The Yesavage Geriatric Depression Scale | Up to twelve weeks
  Questionnaire used to screen for depression in older people. Scores from 00 to 05 indicate Normal screening, 06 to 10 Moderate Depression screening, and 11 to 15 Severe Depression screening.
Anxiety | Up to twelve weeks
  Anxiety was assessed using the Hamilton Scale [25], an instrument designed to identify and measure anxiety symptoms, exploring the alteration of the emotional state, as well as subjective sensations of tension, restlessness or nervousness. The scale consists of 14 items covering physical, mental and behavioural symptoms related to anxiety. Of these items, 7 are aimed at assessing psychological anxiety (items 1-6 and 14), while the other 7 focus on somatic anxiety (items 7-13). Each item is scored on a scale ranging from 0 to 4, where: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe and 4 = Very severe. The total score of the scale ranges from 0 to 56 points, with higher values reflecting a greater intensity of anxiety symptoms.
Perceived Stress | Up to twelve weeks
  The Perceived Stress Scale (PSS) is a self-administered questionnaire designed to measure the level of perceived stress over the past month [28,29]. This instrument consists of 14 items that are answered using a five-point scale (0 = never, 1 = almost never, 2 = sometimes, 3 = often, 4 = very often). To calculate the total score, the responses to items 4, 5, 6, 7, 9, 10, and 13 are reversed (assigning values of 0=4, 1=3, 2=2, 3=1, and 4=0) and then the scores for all items are summed. The total range varies between 0 and 56 points, with higher scores indicating a higher level of perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Paola Romera Gasparico, Jaén, Spain